CLINICAL TRIAL: NCT01188590
Title: Pilot Study: Transcutaneous Carbon Dioxide Monitoring Post Cardiac Surgery: Incidence and Severity of Respiratory Insufficiency
Brief Title: Transcutaneous Carbon Dioxide Monitoring Post Cardiac Surgery: Incidence and Severity Resp Insufficiency
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 009-220
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Respiratory Insufficiency
Keywords: Post operative Respiratory insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing heart surgery
  Interventions: Device: TOSCA 500 monitor

INTERVENTIONS:
Device: TOSCA 500 monitor — transcutaneous ear lobe probe that monitors pulse rate, oxygen saturation and carbon dioxide levels

SUMMARY:
The purpose for the investigators study is to investigate the severity and incidence of respiratory insufficiency using transcutaneous carbon dioxide (TcPCO2) monitoring as an adjunct to the current standard of care for early detection of inadequate ventilation in post-operative surgical in-patients undergoing cardiac surgery after discharge from intensive care unit (ICU) or post anesthesia recovery unit (PACU).

DETAILED DESCRIPTION:
This observational study is to determine the baseline carbon dioxide and severity of respiratory distress and acute respiratory failure (ARF)/respiratory arrest in the post cardiac surgery patients in the first 24 hours on a monitored telemetry floor.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class 1, 2, 3, or 4 men and women who are having cardiac surgery by one of the participating surgeons

Exclusion Criteria:

1. Subject has participated in a trial with any experimental drug or device trial within 30 days prior to enrollment in the study, or has ever been enrolled in this study;
2. Subject has a condition that would require an extensive amount of time off of 13 Roberts during the first 24 hours of admission to the telemetry unit. (e.g., hemodialysis);
3. Subject has a condition or allergy which would prohibit placing the probe on the earlobes;
4. Subject is unable to undergo any procedure required by the protocol;
5. Subject has any other condition or factor which, in the Investigator's opinion, might increase the risk to the subject; or
6. If female, subject is non-lactating, and is either:

   * Not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; or
   * Of childbearing potential but is not pregnant as confirmed by negative serum pregnancy test at time of screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiovascular surgical patients at Baylor University Medical Center
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Determine the baseline TcPCO2 levels for first 24 hours post ICU of cardiac surgery patients. | 24 hours

SECONDARY OUTCOMES:
Classify levels of hypercarbia found | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Ramsay, MD, FRCA, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States